CLINICAL TRIAL: NCT06333353
Title: Is Repetitive Transcranial Magnetic Stimulation Effective in Reducing Endometriosis-associated Pain: A Randomized Controlled Trial
Brief Title: Is Repetitive Transcranial Magnetic Stimulation Effective in Reducing Endometriosis-associated Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Dr. Linda McLean, Professor in the School of Rehabilitation Sciences at University Of Ottawa, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-06-23-9278
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Endometriosis; Pain
Keywords: Repetitive Transcranial Magnetic Stimulation; intervention; endometriosis; pain
MeSH Terms: conditions — Endometriosis; Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, care providers, investigators and outcome assessors will remain blinded to real/sham intervention. The outcomes assessor and the investigator will remain blinded to intervention duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Real RepetitiveTranscranial Magnetic Stimulation (rTMS) 5 sessions (Experimental): The real rTMS intervention will be delivered to the primary motor cortex (M1) on the left side, over the hand representation, using high frequency (HF) rTMS applied by way of a Magstim Rapid² system. The coil position and orientation will be standardized between treatment visits through using a Brainsight neuronavigation system (Rogue Research, Canada). Each of 5 rTMS sessions will consist of a total of 1500 pulses: 15 sets of pulses delivered at 10Hz for 10s at 80% resting motor threshold (RMT), separated by 50s intervals. The real rTMS intervention will be delivered daily over 5 consecutive days.
  Interventions: Device: Real RepetitiveTranscranial Magnetic Stimulation 5 sessions
- Sham RepetitiveTranscranial Magnetic Stimulation (rTMS) 5 sessions (Sham Comparator): The sham rTMS intervention will be delivered to the primary motor cortex (M1) on the left side, over the hand representation, using high frequency (HF) rTMS applied by way of a Magstim Rapid² system interfaced with a placebo coil, whose position and orientation will standardized between treatment visits using a Brainsight neuronavigation system (Rogue Research, Canada) The sham stimulation target will be individually defined at baseline as the site eliciting the highest averaged motor evoked potential (MEP) peak-to-peak amplitude in the first dorsal interosseous (FDI) muscle. Each of 5 sham rTMS sessions will consist of a total of 1500 sham pulses: 15 sets of sham pulses (0% output) delivered at 10Hz for 10s, separated by 50s intervals. The sham intervention will be delivered daily over 5 consecutive days.
  Interventions: Device: Sham RepetitiveTranscranial Magnetic Stimulation 5 sessions
- Real RepetitiveTranscranial Magnetic Stimulation (rTMS) 10 sessions (Experimental): The real 10-session rTMS intervention will be the same as that delivered for the real 5-session rTMS intervention, but delivered as 5 daily sessions, a two day break, and 5 more daily sessions.
  Interventions: Device: Real RepetitiveTranscranial Magnetic Stimulation 10 sessions
- Sham RepetitiveTranscranial Magnetic Stimulation (rTMS) 10 sessions (Sham Comparator): The sham 10 session rTMS intervention will be delivered identically to the sham 5 session intervention, but delivered as 5 daily sessions, a two day break, and 5 more daily sessions.
  Interventions: Device: Sham RepetitiveTranscranial Magnetic Stimulation 10 sessions

INTERVENTIONS:
Device: Real RepetitiveTranscranial Magnetic Stimulation 5 sessions — 5 consecutive treatment sessions will be provided using a protocol based on the updated guideline (Lefaucheur, 2014) and on Pinot-Monange et al. (2019). Each treatment session will last approximately 30 minutes.
  Acceptability, adverse events and side effects will be recorded after each session, while the researchers will also record the total treatment time, difficulties encountered during implementation, and any modifications to the intervention.
  Arms: Real RepetitiveTranscranial Magnetic Stimulation (rTMS) 5 sessions
Device: Sham RepetitiveTranscranial Magnetic Stimulation 5 sessions — 5 consecutive sham treatment sessions will be provided using a protocol based on the updated guideline (Lefaucheur, 2014) and on Pinot-Monange et al. (2019). Each treatment session will last approximately 30 minutes.
  Acceptability, adverse events and side effects will be recorded after each session, while the researchers will also record the total treatment time, difficulties encountered during implementation, and any modifications to the intervention
  Arms: Sham RepetitiveTranscranial Magnetic Stimulation (rTMS) 5 sessions
Device: Real RepetitiveTranscranial Magnetic Stimulation 10 sessions — 10 consective treatment sessions will be provided using a protocol based on the updated guideline (Lefaucheur, 2014) and on Pinot-Monange et al. (2019). Each treatment session will last approximatly 30 minutes.
  Acceptability, adverse events and side effects will be recorded after each session, while the researchers will also record the total treatment time, difficulties encountered during implementation, and any modifications to the intervention.
  Arms: Real RepetitiveTranscranial Magnetic Stimulation (rTMS) 10 sessions
Device: Sham RepetitiveTranscranial Magnetic Stimulation 10 sessions — 10 consective sham treatment sessions will be provided using a protocol based on the updated guideline (Lefaucheur, 2014) and on Pinot-Monange et al. (2019). Each treatment session will last approximatly 30 minutes.
  Acceptability, adverse events and side effects will be recorded after each session, while the researchers will also record the total treatment time, difficulties encountered during implementation, and any modifications to the intervention.
  Arms: Sham RepetitiveTranscranial Magnetic Stimulation (rTMS) 10 sessions

SUMMARY:
The goal of this research is to improve pain outcomes for the over 500K Canadian women, girls and gender-diverse individuals who are newly diagnosed with endometriosis each year. Chronic pain that persists after interventions for endometriosis is a huge problem. There is some evidence that endometriosis-associated pain (EAP) is, at least to some extent, associated with changes in pain physiology, particularly central sensitization of pain. There is currently no effective evidence-informed intervention that addresses EAP. Yet a recent feasibility trial on a repetitive transcranial magnetic stimulation (rTMS) intervention demonstrated promising results compared to a sham intervention for reducing pain in a sample with EAP.

The objectives of this trial are:

1. to evaluate the effectiveness of an rTMS intervention for pain reduction among those with recalcitrant post-operative EAP,
2. to inform on the utility of a long (10 session) vs short (5 session) protocol for pain reduction among those with recalcitrant post-operative EAP
3. to determine if any improvements in pain observed 30 days after an rTMS intervention are retained 6 months later
4. to identify physical and psychosocial mediators that impact the successful reduction of pain among patients with EAP treated using rTMS.
5. to describe patients' perceptions of and satisfaction with rTMS as an intervention for EAP.

DETAILED DESCRIPTION:
This will be a double-blind, randomized-controlled trial (RCT) using a 2X2 factorial design. The protocol was developed following the Consolidated Standards of Reporting Trials (CONSORT) statement and also follows the Canadian Institutes for Health Research (CIHR) Strategy for Patient-Oriented Research (SPOR) to adapt research activities and dissemination strategies to patients equitably and effectively.

The interventions include repetitive transcranial magnetic stimulation (rTMS) delivered using either a real or a sham coil and one of two intervention durations (short: 5-session, long: 10 session), thus four study groups with 1:1:1:1 allocation.

Intervention: The rTMS intervention will be delivered to the primary motor cortex (M1) on the left side, over the hand representation using high frequency (HF) rTMS. Since there is no known somatotopy for pelvic pain, handedness is not thought to be important, however, handedness will be recorded to verify this. The rTMS intervention will be applied by way of a Magstim Rapid² system (Whitland, UK) coupled with a 70mm cooled figure-of-8 coil. The coil position and orientation will be standardized between treatment visits through using a Brainsight neuronavigation system (Rogue Research, Canada). A standard Montreal Neurological Institute (MNI) atlas will be used. The stimulation target will be individually defined at baseline as the site eliciting the highest averaged motor evoked potential (MEP) peak-to-peak amplitude in the first dorsal interosseous (FDI) muscle. The resting motor threshold (RMT) will be defined as the lowest intensity stimulus that elicits a MEP in the FDI of the right hand, with a peak-to-peak amplitude of at least 50 uV in 50% of trials. MEPs will be recorded using the on-board EMG system. Each rTMS session (real or sham) will consist of a total of 1500 pulses: 15 sets of pulses delivered at 10Hz for 10s at 80% RMT, separated by 50s intervals. The short protocol will involve interventions on 5 consecutive days, while the long protocol will include a 2-day break and another 5- day intervention. Acceptability, adverse events and side effects will be recorded after each session. Missed visits will be rescheduled wherever possible (but tracked). and adherence will be recorded as a proportion of sessions attended.

Participant allocation: Concealed, computer-generated allocation will be performed using permuted block randomization (block size= 4) only after a participant has consented and completed all questionnaires at baseline. The allocation sequence will be managed by an independent investigator not associated with the project. It will be concealed from the study team through storage in a password protected file on an encrypted computer, backed up in a password-protected directory. Groups will be labelled as A-short, A-long, B-short, B-long, to keep investigators and participants blinded as to which coil (A/B) provides real/sham rTMS (only one investigator who will have no direct involvement with participants will know which coil provides real/sham rTMS; they look, sound and feel identical). Treatment duration will be revealed only to the recruitment officer, to the individual delivering the intervention, and the participant, since they will need to know the length of the protocol to schedule intervention sessions and follow-up. Gender will be recorded and if possible, gender-based sub-analyses will be performed. the sample will not be stratified by race/ethnicity, however efforts will be made to ensure diversity in the sample, as the prevalence of endometriosis also appears to be influenced by race/ethnicity. Recruitment bias will be minimized through using multiple recruitment sources with broad reach. Consistent with the CONSORT extension recommendations for trials involving non-pharmacological interventions, the researchers who perform baseline and follow-up assessments will not be involved in the treatment, and will be blinded to group allocation.

Data collection: A series of questionnaires will be completed using an on-line platform before and after the intervention and laboratory-based assessments will occur on the day of the first and final (5th or 10th) intervention session, at the later of which participants will report their patient global impression of change (PGIC) in pain, and their patient satisfaction with treatment (PST). All participants will be followed daily to record their daily pain (NRS 0-10) in the 30 days before the first and 30 days after the last rTMS intervention session using automated text messaging or e-mail notifications, or phone calls if that is their preference. 30 days after the intervention (primary end point), and 6 months later, participants will provide their PGIC for pain, PST, and complete the Brief Pain inventory (BPI), the Endometriosis Health Profile (EHP-30) and the Beck Depression Index (BDI), through an on-line platform (reminders will be sent and non-completion will be monitored, with follow-up by the protocol officer to ensure completion wherever possible). Individuals randomized to the real intervention (both short and long protocols) will be invited to participate in a semi-structured interview through which we aim to capture a nuanced impression of the effectiveness of the intervention, its acceptability, and other observations.

Target Sample size: The target sample size is 152 participants (38 per group). The sample size was estimated based on findings of a prospective cohort study by Pinot-Monange et al. which suggested that 75% of participants (9 of 12) will be improved on the PGIC, and that there will be a reduction in reported pain sensitivity (d=0.62) associated with the short rTMS protocol. The rTMS literature suggests that a moderate effect size (Cohen's d=0.05), will be achieved, suggesting that a sample of 30 per group will provide sufficient power to detect an intervention effect. A simulation in R based on 100 replications using a small (d=0.2) effect suggested that such an interaction would be detected (power = 0.80) with a sample size of n=100 (25 per group). The sample size includes estimated conservative drop-out rates, 15%, at the primary end point, and 25% after 6 months.

Recruitment sources: Recruitment will be from a broad range of sources within the Ottawa, Ontario and Gatineau Quebec regions of Canada, including local gynecology clinics, local physiotherapy clinics, social media platforms (Instagram, X, Facebook), printed posters at sites within the community related to social interests, cultural practices, and religious beliefs, and sexual health resource centers.

Planned analyses: Baseline participant characteristics will be aggregated by group and summarized using descriptive statistics. Intent-to-treat analyses will be performed to address Objectives 1-3. To answer Objectives 1 and 2, and to address relevant secondary objectives, 2-way repeated-measures ANOVAs will be performed for continuous variables, including intervention (2 levels: real, sham) and duration (2 levels: short, long) as main effects, and the interaction between intervention and duration, using α=0.05 and adjusting for unequal variances if necessary. Where there are significant interaction effects, Cohen's d and marginal means will be used to estimate effect sizes. Where no significant interactions are found, within- and between-group main effects will be estimated using Cohen's d. Chi-Square analyses will be used to evaluate group differences in the proportion of participants reporting meaningful clinical changes in pain based on the average daily pain (>30% improvement) and the PGIC (somewhat to very much improved), generating Odds Ratios and estimating the number needed to treat with 95% confidence. Analyses after the 6- month follow-up will include time as a main effect. Wherever possible, the data will be disaggregated by gender and race/ethnicity, and sub-analyses will be performed. Where this is not possible, descriptive analyses by gender and race/ethnicity will be reported, highlighting observations that may inform future studies.

To address Objective 4, univariate analyses using only data from those who received real rTMS will be used to identify trends (p<0.15) in baseline and demographic data such as, age, race, gender, daily pain, EHP-30, BPI, Central Sensitization Inventory (CSI), Pain Catastrophizing Scale (PCS), BDI, State Trait Anxiety Inventory (STAI), pressure pain threshold (PPThresh), pressure pain tolerance (PPTol), temporal summation of pain (TS), conditioned pain modulation (CPM) and Tampon Test, suggestive of differences between successes (>30% improvement) and failures. Separate binary logistic regression models will examine the relationship between independent variables tending to differ by group and clinically relevant improvements in dependent variables [PGIC (somewhat to very much improved), daily pain (>30% improved), BPI (> 30% improved) and EHP-30(> 30% improved). Only three predictors will be included in the final model- the one's with the largest effect sizes in univariate testing. Bootstrapping (X1000) will be used to improve the robustness of the models.

Recruitment rate, adherence, adverse events and use of rescue medications (reported on the BPI) will be analyzed descriptively, and any protocol deviations will be described. Post-intervention interview data will be coded, and a thematic analysis will be completed in duplicate using N-Vivo software. Interviews will continue until 15 have been completed, thematic saturation is reached, and no new themes emerge after three consecutive interviews.

Planned Interim analyses: One interim analysis will be performed once n=16 per group have reached the primary endpoint and based on Question 1. The trial will be deemed futile if the conditional power to detect a treatment effect for all intervention groups is <30%. The trial will not be deemed futile based on the power of the interaction effect.

ELIGIBILITY:
Inclusion Criteria:

-self-reported endometriosis-associated pain (> 3 in the numeric rating scale, 0-10) that has persisted following medical or surgical intervention,

Exclusion Criteria:

* Contra-indications to rTMS (e.g., metal/implants around the head/neck, pacemaker), history of epilepsy (history of seizures) in the family
* Pain symptoms initiated by other known causes (e.g., infections, thyroid disease, autoimmune diseases, gastrointestinal disease)
* Experience a more severe, extra-pelvic pain than that associated with endometriosis
* Pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) used to record daily pain over 30 days | Baseline -30 days after enrolment and before allocation
  Pain intensity, using a numeric rating scale (NRS), will be recorded daily for 30 days prior to trial entry to provide a suitable baseline,
  It will measure the average and worst overall pain intensity, menstrual and sexual activity related pain (if applicable).
  The questions will be applied as described below:
  Please rate any pain you experienced today (over the past 24 hours) that you attribute to your endometriosis using a scale from 0 (no pain) to 10 (worst pain imaginable).
  Is today your first day of menstrual cycle?
  Did you attempt any sexual activity or tampon insertion in the last 24hs? Please rate the pain associated with this activity on a scale from 0 (no pain) to 10 (worst pain imaginable),for sexual activity and/or tampon insertion (if applicable).
Numeric rating scale(NRS) used to record daily pain over 30 days | 30 days following intervention
  Pain intensity, using a numeric rating scale (NRS), will be recorded daily after the intervention period for 30 days.
  It will measure the average and worst overall pain intensity, menstrual and sexual activity related pain (if applicable).
  The questions will be applied as described below:
  Please rate any pain you experienced today (over the past 24 hours) that you attribute to your endometriosis using a scale from 0 (no pain) to 10 (worst pain imaginable).
  Is today your first day of menstrual cycle?
  Did you attempt any sexual activity or tampon insertion in the last 24hs? Please rate the pain associated with this activity on a scale from 0 (no pain) to 10 (worst pain imaginable), for sexual activity and/or tampon insertion (if applicable).
Patient Global Impression of Change (PGIC) in pain | After the Intervention on the final intervention day
  PGIC is a single question through which participants provide a ordinal rating based on their overall perception of change in their pain attributed to the intervention:
  Very Much Better, Much Better, Somewhat better, About the same, somewhat worse, much worse, very much worse
Patient Global Impression of Change (PGIC) in pain | 30 days after completing the intervention
  PGIC is a single question through which participants provide a ordinal rating based on their overall perception of change in their pain attributed to the intervention:
  Very Much Better, Much Better, Somewhat better, About the same, somewhat worse, much worse, very much worse
Patient Global Impression of Change (PGIC) in pain | 6 months after the intervention
  PGIC is a single question through which participants provide a ordinal rating based on their overall perception of change in their pain attributed to the intervention:
  Very Much Better, Much Better, Somewhat better, About the same, somewhat worse, much worse, very much worse

SECONDARY OUTCOMES:
The Beck Depression Inventory (BDI-II) | Baseline
  The 21-item self-administered survey is scored on a scale of 0-3 in a list of four statements arranged in increasing severity about a symptom of depression. BDI-II assesses presence and intensity of mood symptoms. The scale can be divided into 2 subscales, affective symptoms (8 items) and somatic symptoms (13 items). Cut-off scores are available to classify degree of mood intensity.
  There is a four-point scale for each item ranging from 0 to 3. On two items (16 and 18) there are seven options to indicate either an increase or decrease of appetite and sleep. Cut-off score guidelines for the BDI-II are given with the recommendation that thresholds be adjusted based on the characteristics of the sample, and the purpose for use of the BDI-II. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe. This scale can be scored either manually or using the Pearson proprietary software Q-global.
The Beck Depression Inventory (BDI-II) | 30 days following the intervention
  The 21-item self-administered survey is scored on a scale of 0-3 in a list of four statements arranged in increasing severity about a symptom of depression. BDI-II assesses presence and intensity of mood symptoms. The scale can be divided into 2 subscales, affective symptoms (8 items) and somatic symptoms (13 items). Cut-off scores are available to classify degree of mood intensity.
  There is a four-point scale for each item ranging from 0 to 3. On two items (16 and 18) there are seven options to indicate either an increase or decrease of appetite and sleep. Cut-off score guidelines for the BDI-II are given with the recommendation that thresholds be adjusted based on the characteristics of the sample, and the purpose for use of the BDI-II. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe. This scale can be scored either manually or using the Pearson proprietary software Q-global.
The Beck Depression Inventory (BDI-II) | 6 months following the intervention
  The 21-item self-administered survey is scored on a scale of 0-3 in a list of four statements arranged in increasing severity about a symptom of depression. BDI-II assesses presence and intensity of mood symptoms. The scale can be divided into 2 subscales, affective symptoms (8 items) and somatic symptoms (13 items). Cut-off scores are available to classify degree of mood intensity.
  There is a four-point scale for each item ranging from 0 to 3. On two items (16 and 18) there are seven options to indicate either an increase or decrease of appetite and sleep. Cut-off score guidelines for the BDI-II are given with the recommendation that thresholds be adjusted based on the characteristics of the sample, and the purpose for use of the BDI-II. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe. This scale can be scored either manually or using the Pearson proprietary software Q-global.
The State-Trait Anxiety Inventory (STAI) | Baseline
  The State-Trait Anxiety Inventory (STAI) (Stauder, 2003) allows discrimination between anxiety as a personality trait (STAI-T) or as an emotional response to a situation (STAI-S). This 40-item scale has shown a good reliability, consistency, and responsiveness (Sepulcri, 2009). Using the STAI, Sepulcri & do Amaral (Sepulcri, 2009) reported that 87.5% of patients with EAP reported anxiety, with significant associations between both STAI-T and STAI-S and pain intensity.
  Total scores for state and trait are calculated, ranging from 20 - 80. Higher scores indicate greater anxiety.
  1. = Scores between 20-39 means "no or low anxiety"
  2. = Scores between 40-59 means "moderate anxiety"
  3. = Scores between 60-80 means "high anxiety"
The Pain Catastrophizing Scale | Baseline
  This is a reliable and valid scale to measure of catastrophizing. The scores from this questionnaire is predictors of intensity of physical and emotional distress. It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present.
The Central sensitization index | Baseline
  The Central Sensitisation Inventory (CSI) is a self-report outcome measure designed to identify patients who have symptoms that may be related to central sensitisation (CS) or central sensitivity syndromes (CSS). Part A includes 25 questions related to common CSS symptoms.
  Part B determines if the patient has been diagnosed with certain CSS disorders or related disorders, such as anxiety and depression. CSI severity levels have been established for part A: subclinical = 0 to 29; mild = 30 to 39; moderate = 40 to 49; severe = 50 to 59; and extreme = 60 to 100.
Female Sexual Distress Scale (FSDS) | Baseline
  The Female Sexual Distress Scale-Revised (FSDS-R) is a 13-item questionnaire designed to assess sexually related distress in women with hypoactive sexual desire disorder (HSDD). It has been validated for evaluating distress associated with inadequate or impaired sexual function.
  The total score on the FSDS-R ranges from 0 to 48, with higher scores indicating higher levels of sexual distress. A cutoff score of 15 or more is recommended for determining the presence of personal sexual distress.
Adherence to the intervention protocol | During intervention sessions
  Attendance of rTMS treatment visits will be tracked (%).
Pressure pain threshold (PPThresh) | Baseline before allocation
  PPT will be determined using an algometer device in three regions over the lower abdomen [lower left and right quadrants (4cm medial to the anterior superior iliac spine) and midline (1 cm superior to the midline pubic symphysis)]. Three sites remote to the pelvis (right thenar eminence, right upper trapezius, and right medial gastrocnemius) will also be assessed.
  PPT will be defined as the median pressure (Newton), among three trials, at which participants first report pain.
  After each pressure application participants will be asked to rate their pain using the NRS from 0 to 10.
Pressure pain threshold (PPThresh) | After the final intervention session on the same day as that session
  PPT will be determined using an algometer device in three regions over the lower abdomen [lower left and right quadrants (4cm medial to the anterior superior iliac spine) and midline (1 cm superior to the midline pubic symphysis)]. Three sites remote to the pelvis (right thenar eminence, right upper trapezius, and right medial gastrocnemius) will also be assessed.
  PPT will be defined as the median pressure (Newton), among three trials, at which participants first report pain.
  After each pressure application participants will be asked to rate their pain using the NRS from 0 to 10.
Pressure Pain Tolerance (PPTol) | Baseline before allocation
  PPTol will be determined using an algometer device in three regions over the lower abdomen [lower left and right quadrants (4cm medial to the anterior superior iliac spine) and midline (1 cm superior to the midline pubic symphysis)]. Three sites remote to the pelvis (right thenar eminence, right upper trapezius, and right medial gastrocnemius) will also be assessed.
  PPTol will be defined as the median pressure (Newton), among three trials, at which participants can tolerate the pressure before the sensation becomes intolerable or unbearable.
  After each pressure application participants will be asked to rate their pain in a numerical rating scale (NRS) from 0 to 10.
Pressure Pain Tolerance (PPTol) | Immediately after the final intervention session
  PPTol will be determined using an algometer device in three regions over the lower abdomen [lower left and right quadrants (4cm medial to the anterior superior iliac spine) and midline (1 cm superior to the midline pubic symphysis)]. Three sites remote to the pelvis (right thenar eminence, right upper trapezius, and right medial gastrocnemius) will also be assessed.
  PPTol will be defined as the median pressure (Newton), among three trials, at which participants can tolerate the pressure before the sensation becomes intolerable or unbearable.
  After each pressure application participants will be asked to rate their pain in a numerical rating scale (NRS) from 0 to 10.
Perceived pain intensity (PPI) | Baseline before allocation
  Perceived pain intensity (PPI) will be applied, using an algometer device during 5 seconds using the mean pressure between PPThresh and PPTol obtained previously for each participant, in all sites described above. After each pressure application participants will be asked to rate their pain in a numerical rating scale (NRS) from 0 to 10.
Perceived pain intensity (PPI) | Immediately after the final intervention session
  Perceived pain intensity (PPI) will be applied, using an algometer device during 5 seconds using the mean pressure between PPThresh and PPTol obtained previously for each participant, in all sites described above. After each pressure application participants will be asked to rate their pain in a numerical rating scale (NRS) from 0 to 10.
Temporal summation (TS) of pain | Baseline before allocation
  TS is reflective of sensitization through peripheral and/or central mechanisms. The stimulus intensity will be the PPI determined above at the midline lower abdominal site and at the thenar site, determined during pressure pain threshold (PPT) assessment. Ten stimuli will be delivered at each site at a rate of one per second. Pain intensity reported using a NRS, induced by the application of the stimulus on the 1st and 10th application will be recorded. TS will be considered as a dichotomous variable, deemed to be present if there is a positive difference > 1 between NRS ratings on the tenth minus that of the first application of the stimulus and negative otherwise
Temporal summation (TS) of pain | Immediately after the final intervention session
  TS is reflective of sensitization through peripheral and/or central mechanisms. The stimulus intensity will be the PPI at the lower abdominal site and at the thenar site, determined during pressure pain threshold (PPT) assessment. Ten stimuli will be delivered at each site at a rate of one per second. Pain intensity reported using a NRS, induced by the application of the stimulus on the 1st and 10th application will be recorded. TS will be considered as a dichotomous variable, deemed to be present if there is a positive difference > 1 between NRS ratings on the tenth minus that of the first application of the stimulus and negative otherwise
Pain rating during the tampon test | Baseline before allocation
  The participants will be provided with Original Regular Tampax Tampon and will be instructed to insert and then remove it. After, they will be asked to record the degree of pain during the entire insertion/removal experience in a 11-point numerical rating scale (NRS) with anchors of 0 (no pain at all) to 10 (worst pain imaginable).
Pain rating during the tampon test | Immediately after the final intervention session
  The participants will be provided with Original Regular Tampax Tampon and will be instructed to insert and then remove it. After, they will be asked to record the degree of pain during the entire insertion/removal experience in a 11-point numerical rating scale (NRS) with anchors of 0 (no pain at all) to 10 (worst pain imaginable).
Conditioned pain modulation (CPM) | Baseline before allocation
  CPM is manifested by a reduction in pain perception in one location through the simultaneous application of a painful stimulus at a distant, non-segmental location on the body. A lack of CPM is reflective of decreased descending endogenous pain inhibition, a contributor to central sensitization.
  Through the PPThresh (test stimulus) will be tested at the lower midline abdominal site and the thenar eminence site. A blood pressure cuff will be applied to the dominant upper arm and inflated at a rate of 20 mmHg/s until the participant reports a pain intensity of 3/10 (conditioning stimulus). The test stimulus will be repeated 3X at each site while the pressure is retained at the upper arm. CPM will be deemed present if the median PPThresh is lower with the conditioning stimulus applied than prior to the conditioning stimulus.
Conditioned pain modulation (CPM) | Immediately after the final intervention session
  CPM is manifested by a reduction in pain perception in one location through the simultaneous application of a painful stimulus at a distant, non-segmental location on the body. A lack of CPM is reflective of decreased descending endogenous pain inhibition, a contributor to central sensitization.
  Through the PPThresh (test stimulus) will be tested at the lower midline abdominal site and the thenar eminence site. A blood pressure cuff will be applied to the dominant upper arm and inflated at a rate of 20 mmHg/s until the participant reports a pain intensity of 3/10 (conditioning stimulus). The test stimulus will be repeated 3X at each site while the pressure is retained at the upper arm. CPM will be deemed present if the median PPThresh is lower with the conditioning stimulus applied than prior to the conditioning stimulus.
The Brief Pain Inventory | Baseline before allocation
  It evaluates a patient's pain experience over the previous 1 weeks through locating the pain, noting medication or other interventions, and 11 different numeric rating scales (NRSs) ask about pain intensity (current, least, most, and average for the past 24 hours) and the effect of the pain on function during various activities of daily living. The BPI is an excellent tool for monitoring the effect of pain or treatment of pain, or both, in terms of a patient's functional ability or disability over time. Cronbach alpha reliability ranges from 0.77 to 0.91.
  Scoring: The short version of the BPI (Short form) includes 9 items. It uses a 0 to 10 numeric rating scales for item rating.
  Pain Score:
  * 1 - 4 = Mild Pain
  * 5 - 6 = Moderate Pain
  * 7 - 10 = Severe Pain
The Brief Pain Inventory | 30 days after the final intervention session
  It evaluates a patient's pain experience over the previous 7 days through locating the pain, noting medication or other interventions, and 11 different numeric rating scales (NRSs) ask about pain intensity (current, least, most, and average for the past 24 hours) and the effect of the pain on function during various activities of daily living. The BPI is an excellent tool for monitoring the effect of pain or treatment of pain, or both, in terms of a patient's functional ability or disability over time. Cronbach alpha reliability ranges from 0.77 to 0.91.
  Scoring: The short version of the BPI (Short form) includes 9 items. It uses a 0 to 10 numeric rating scales for item rating.
  Pain Score:
  * 1 - 4 = Mild Pain
  * 5 - 6 = Moderate Pain
  * 7 - 10 = Severe Pain
The Brief Pain Inventory | 6 months after the final intervention session
  It evaluates a patient's pain experience over the previous 1 weeks through locating the pain, noting medication or other interventions, and 11 different numeric rating scales (NRSs) ask about pain intensity (current, least, most, and average for the past 24 hours) and the effect of the pain on function during various activities of daily living. The BPI is an excellent tool for monitoring the effect of pain or treatment of pain, or both, in terms of a patient's functional ability or disability over time. Cronbach alpha reliability ranges from 0.77 to 0.91.
  Scoring: The short version of the BPI (Short form) includes 9 items. It uses a 0 to 10 numeric rating scales for item rating.
  Pain Score:
  * 1 - 4 = Mild Pain
  * 5 - 6 = Moderate Pain
  * 7 - 10 = Severe Pain
The Endometriosis Health Profile Questionnaire (EPH-30) | Baseline before allocation
  The 30 questions of the EHP-30 involve five scales (pain, control and powerlessness, emotional well-being, social support, and self-image) answered based on a 4-week recall period. Higher scores (/100) reflect better health.
The Endometriosis Health Profile Questionnaire (EPH-30) | 30 days after the final intervention session
  The 30 questions of the EHP-30 involve five scales (pain, control and powerlessness, emotional well-being, social support, and self-image) answered based on a 4-week recall period. Higher scores (/100) reflect better health.
The Endometriosis Health Profile Questionnaire (EPH-30) | 6 months after the final intervention session
  The 30 questions of the EHP-30 involve five scales (pain, control and powerlessness, emotional well-being, social support, and self-image) answered based on a 4-week recall period. Higher scores (/100) reflect better health.
Patient satisfaction with treatment (PST) | Immediately after the intervention on the final day of the intervention
  Global patient satisfaction with treatment is a single question through which participants provide their rating of satisfaction using a scale from zero to ten. Higher ratings reflect greater satisfaction.
Patient satisfaction with treatment (PST) | 30 days after the final intervention session
  Global patient satisfaction with treatment is a single question through which participants provide their rating of satisfaction using a scale from zero to ten. Higher ratings reflect greater satisfaction.
Patient satisfaction with treatment (PST) | 6 months after the final intervention session
  Global patient satisfaction with treatment is a single question through which participants provide their rating of satisfaction using a scale from zero to ten. Higher ratings reflect greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Linda McLean, PhD, Principal Investigator — University of Ottawa
Locations (1):
- McLean Function Measurement Lab, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Spreadsheets will be provide by email upon request and based on the planned use of the data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 10 years after the publication of the study results
Access Criteria: Planned use of data for systematic review or meta-analysis.

REFERENCES:
- [Background] Bajaj P, Bajaj P, Madsen H, Arendt-Nielsen L. Endometriosis is associated with central sensitization: a psychophysical controlled study. J Pain. 2003 Sep;4(7):372-80. doi: 10.1016/s1526-5900(03)00720-x. PMID 14622679
- [Background] Gatchel RJ, Peng YB, Peters ML, Fuchs PN, Turk DC. The biopsychosocial approach to chronic pain: scientific advances and future directions. Psychol Bull. 2007 Jul;133(4):581-624. doi: 10.1037/0033-2909.133.4.581. PMID 17592957
- [Background] Kennedy DL, Kemp HI, Ridout D, Yarnitsky D, Rice ASC. Reliability of conditioned pain modulation: a systematic review. Pain. 2016 Nov;157(11):2410-2419. doi: 10.1097/j.pain.0000000000000689. PMID 27559835
- [Background] O'Connell NE, Marston L, Spencer S, DeSouza LH, Wand BM. Non-invasive brain stimulation techniques for chronic pain. Cochrane Database Syst Rev. 2018 Mar 16;3(3):CD008208. doi: 10.1002/14651858.CD008208.pub4. PMID 29547226
- [Background] Singh S, Soliman AM, Rahal Y, Robert C, Defoy I, Nisbet P, Leyland N. Prevalence, Symptomatic Burden, and Diagnosis of Endometriosis in Canada: Cross-Sectional Survey of 30 000 Women. J Obstet Gynaecol Can. 2020 Jul;42(7):829-838. doi: 10.1016/j.jogc.2019.10.038. Epub 2020 Jan 27. PMID 32001176
- [Background] McNamara HC, Frawley HC, Donoghue JF, Readman E, Healey M, Ellett L, Reddington C, Hicks LJ, Harlow K, Rogers PAW, Cheng C. Peripheral, Central, and Cross Sensitization in Endometriosis-Associated Pain and Comorbid Pain Syndromes. Front Reprod Health. 2021 Sep 1;3:729642. doi: 10.3389/frph.2021.729642. eCollection 2021. PMID 36303969
- [Background] Carey ET, Martin CE, Siedhoff MT, Bair ED, As-Sanie S. Biopsychosocial correlates of persistent postsurgical pain in women with endometriosis. Int J Gynaecol Obstet. 2014 Feb;124(2):169-73. doi: 10.1016/j.ijgo.2013.07.033. Epub 2013 Oct 31. PMID 24290537
- [Background] Coccia ME, Rizzello F, Palagiano A, Scarselli G. Long-term follow-up after laparoscopic treatment for endometriosis: multivariate analysis of predictive factors for recurrence of endometriotic lesions and pain. Eur J Obstet Gynecol Reprod Biol. 2011 Jul;157(1):78-83. doi: 10.1016/j.ejogrb.2011.02.008. Epub 2011 Apr 9. PMID 21481523
- [Background] Pagano RL, Fonoff ET, Dale CS, Ballester G, Teixeira MJ, Britto LRG. Motor cortex stimulation inhibits thalamic sensory neurons and enhances activity of PAG neurons: possible pathways for antinociception. Pain. 2012 Dec;153(12):2359-2369. doi: 10.1016/j.pain.2012.08.002. Epub 2012 Sep 25. PMID 23017297
- [Background] Leung A, Donohue M, Xu R, Lee R, Lefaucheur JP, Khedr EM, Saitoh Y, Andre-Obadia N, Rollnik J, Wallace M, Chen R. rTMS for suppressing neuropathic pain: a meta-analysis. J Pain. 2009 Dec;10(12):1205-16. doi: 10.1016/j.jpain.2009.03.010. Epub 2009 May 23. PMID 19464959
- [Background] Pinot-Monange A, Moisset X, Chauvet P, Gremeau AS, Comptour A, Canis M, Pereira B, Bourdel N. Repetitive Transcranial Magnetic Stimulation Therapy (rTMS) for Endometriosis Patients with Refractory Pelvic Chronic Pain: A Pilot Study. J Clin Med. 2019 Apr 13;8(4):508. doi: 10.3390/jcm8040508. PMID 31013910
- [Background] Turk DC, Dworkin RH, Burke LB, Gershon R, Rothman M, Scott J, Allen RR, Atkinson HJ, Chandler J, Cleeland C, Cowan P, Dimitrova R, Dionne R, Farrar JT, Haythornthwaite JA, Hertz S, Jadad AR, Jensen MP, Kellstein D, Kerns RD, Manning DC, Martin S, Max MB, McDermott MP, McGrath P, Moulin DE, Nurmikko T, Quessy S, Raja S, Rappaport BA, Rauschkolb C, Robinson JP, Royal MA, Simon L, Stauffer JW, Stucki G, Tollett J, von Stein T, Wallace MS, Wernicke J, White RE, Williams AC, Witter J, Wyrwich KW. Developing patient-reported outcome measures for pain clinical trials: IMMPACT recommendations. Pain. 2006 Dec 5;125(3):208-215. doi: 10.1016/j.pain.2006.09.028. Epub 2006 Oct 25. No abstract available. PMID 17069973
- [Background] Neelakantan D, Omojole F, Clark TJ, Gupta JK, Khan KS. Quality of life instruments in studies of chronic pelvic pain: a systematic review. J Obstet Gynaecol. 2004 Nov;24(8):851-8. doi: 10.1080/01443610400019138. PMID 16147635
- [Background] Jones G, Kennedy S, Barnard A, Wong J, Jenkinson C. Development of an endometriosis quality-of-life instrument: The Endometriosis Health Profile-30. Obstet Gynecol. 2001 Aug;98(2):258-64. doi: 10.1016/s0029-7844(01)01433-8. PMID 11506842
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Bourdel N, Alves J, Pickering G, Ramilo I, Roman H, Canis M. Systematic review of endometriosis pain assessment: how to choose a scale? Hum Reprod Update. 2015 Jan-Feb;21(1):136-52. doi: 10.1093/humupd/dmu046. Epub 2014 Sep 1. PMID 25180023
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Background] Neblett R, Cohen H, Choi Y, Hartzell MM, Williams M, Mayer TG, Gatchel RJ. The Central Sensitization Inventory (CSI): establishing clinically significant values for identifying central sensitivity syndromes in an outpatient chronic pain sample. J Pain. 2013 May;14(5):438-45. doi: 10.1016/j.jpain.2012.11.012. Epub 2013 Mar 13. PMID 23490634
- [Background] Orr NL, Wahl KJ, Lisonek M, Joannou A, Noga H, Albert A, Bedaiwy MA, Williams C, Allaire C, Yong PJ. Central sensitization inventory in endometriosis. Pain. 2022 Feb 1;163(2):e234-e245. doi: 10.1097/j.pain.0000000000002351. PMID 34030173
- [Background] Sepulcri Rde P, do Amaral VF. Depressive symptoms, anxiety, and quality of life in women with pelvic endometriosis. Eur J Obstet Gynecol Reprod Biol. 2009 Jan;142(1):53-6. doi: 10.1016/j.ejogrb.2008.09.003. Epub 2008 Nov 17. PMID 19010584
- [Background] Morin M, Morin A, Gougeon V, Marchand S, Waddell G, Bureau YA, Girard I, Brassard A, Benoit-Piau J, Leonard G. Transcranial direct current stimulation for provoked vestibulodynia: What roles do psychosexual factors play in treatment response? J Clin Neurosci. 2021 Nov;93:54-60. doi: 10.1016/j.jocn.2021.08.003. Epub 2021 Sep 11. PMID 34656261
- [Background] Stratton P, Khachikyan I, Sinaii N, Ortiz R, Shah J. Association of chronic pelvic pain and endometriosis with signs of sensitization and myofascial pain. Obstet Gynecol. 2015 Mar;125(3):719-728. doi: 10.1097/AOG.0000000000000663. PMID 25730237
- [Background] McLean L, Charette M, Varette K, Brooks K, Harvey MA, Robert M, Baker K, Day A, Della Zazzera V, Sauerbrei E, Brison R. Pelvic floor muscle training as an adjunct to a midurethral sling: a single-blind randomised controlled trial. Int Urogynecol J. 2022 Apr;33(4):809-819. doi: 10.1007/s00192-020-04668-9. Epub 2021 Mar 3. PMID 33660001
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491